CLINICAL TRIAL: NCT02459483
Title: Evaluation of a Telephone Care Nurse in the Management of Patients With Cancer and Treated by Oral Chemotherapy
Acronym: ETICCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut de Cancérologie de la Loire (Other)
Collaborators: Hôpital Privé de la Loire (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-01
Record Dates: First submitted 2015-05-29; First posted 2015-06-02 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nurse phone call (Experimental): a nurse will interview patients by phone every 14 +/- 2 days for 6 months
  Interventions: Behavioral: Nurse phone call
- Control Group (No Intervention): Common practice

INTERVENTIONS:
Behavioral: Nurse phone call
  Arms: Nurse phone call

SUMMARY:
The purpose of this study is to assess the effectiveness of a nurse telephone interview in the management of cancer patients treated by oral chemotherapy. This is a multicenter prospective randomized controlled pragmatic interventional trial conducted in collaboration with two oncology care facilities. Eligible population consists of all patients suffering from advanced cancer and treated by oral chemotherapy except hormonotherapy. 184 patients will be enrolled in the study. The experimental group will receive a standard followed by a medical oncologist, hematologist or radiation therapist as part of routine care, and telephone interviews by a nurse every 14 +/- 2 days for 6 months. The control group will receive a standard followed by a medical oncologist, hematologist or radiation therapist as part of routine care.

The effectiveness of the intervention will be evaluated by a toxicity score of the 9 most common side effects of oral cancer (oral mucositis, hand-foot syndrome, diarrhea, nausea, vomiting, pain, asthenia, rash and anorexia) officers from NCI CTCAE v4.0-(Common Toxicity Criteria for Adverse Events) and turned into a single composite criterion (sum of 9 Toxicity grades).

ELIGIBILITY:
Inclusion Criteria:

* aged over 18 years
* treated in medical oncology, hematology or radiotherapy
* to receive any oral chemotherapy for any cancer except hormone therapy according to decision of the Meeting of Consultation Multidisciplinary

Exclusion Criteria:

* Refusal of participation, protected adult patient under guardianship.
* Patient currently treated with oral chemotherapy
* Patient already included in another clinical research protocol including telephone follow-up
* Patient followed by a Nurse navigators or participating in a therapeutic education program
* Patient concomitantly treated with an injectable chemotherapy regimen or radiotherapy unless irradiation palliative analgesic.
* Patient in inability to understand how the study or inability to follow a telephone conversation.
* Patient with documented history of cognitive or psychiatric disorders.
* Patient residing outside the Rhône Alpes area
* Patient doesn't understand French
* Patient with no phone means

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-11 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Toxicity score | 6 months
  Toxicity Score 9 most common side effects of oral chemotherapy (oral mucositis, hand-foot syndrome, diarrhea, nausea, vomiting, pain, asthenia, rash and anorexia) officers from the NCI-CTCAE v4.0 (Common Toxicity Criteria for Adverse Events) and turned into a single composite criterion (sum of 9 toxicity grades)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hopital Privé de la Loire, Saint-Etienne
  - Institut de Cancerologie de la Loire, Saint-Priest-en-Jarez

REFERENCES:
- [Derived] Bouleftour W, Muron T, Guillot A, Tinquaut F, Rivoirard R, Jacquin JP, Saban-Roche L, Boussoualim K, Tavernier E, Augeul-Meunier K, Collard O, Mery B, Pupier S, Oriol M, Bourmaud A, Fournel P, Vassal C. Effectiveness of a nurse-led telephone follow-up in the therapeutic management of patients receiving oral antineoplastic agents: a randomized, multicenter controlled trial (ETICCO study). Support Care Cancer. 2021 Aug;29(8):4257-4267. doi: 10.1007/s00520-020-05955-3. Epub 2021 Jan 7. PMID 33409726